CLINICAL TRIAL: NCT04757116
Title: A Post-Market, Prospective, Randomized, Controlled, Multicenter International Study to Assess the Safety of the Temporarily Implanted Nitinol Device (iTind) Compared to the UroLift® System in Subjects With Symptomatic Benign Prostatic Hyperplasia (BPH)
Brief Title: Post-Market Study to Assess iTind Safety in Comparison to UroLift
Acronym: MT-08
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Corporation of the Americas (Industry)
Collaborators: Olympus Europe SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT-08
Record Dates: First submitted 2021-02-07; First posted 2021-02-17 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iTind arm (Experimental): The iTind is a minimally invasive temporary implant
  Interventions: Device: iTind
- UroLift (Active Comparator): The UroLift is a minimally invasive permanent implant
  Interventions: Procedure: UroLift

INTERVENTIONS:
Device: iTind — The iTind is implemented for 5-7 days
  Arms: iTind arm
Procedure: UroLift — UroLift is a minimally invasive procedure where permanent implants are placed in the prostate.
  Arms: UroLift

SUMMARY:
The study objective is to evaluate the safety of the iTind device comparied to UroLift.

DETAILED DESCRIPTION:
Both iTind and UroLift are minimally invasive treatment options for relieving lower urinary tract symptoms (LUTS) secondary to benign prostatic hyperplasia (BPH). The iTind device is a temporary, self-expanding nitinol implant that remains in place for 5 to 7 days to reshape the prostatic urethra through localized ischemic pressure and tissue remodeling. In contrast, the UroLift system involves the permanent placement of transprostatic implants that retract the enlarged lateral lobes of the prostate to widen the urethral lumen.

This study is designed to directly compare the safety and effectiveness of the iTind device versus the UroLift system in treating LUTS due to BPH.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of lower urinary tract symptoms presumed to be secondary to benign prostatic enlargement causing bladder outlet obstruction for which treatment is recommended
2. Willing and able to provide informed consent
3. Males ≥ 50 years of age or older
4. PSA < 4 ng/dl, ng/ml or if the PSA is 4 - 10 ng/dl, ng/ml, prostate cancer must be ruled out to the satisfaction of the Principal Investigator (PI) by local standard of care methods within prior 6 months
5. Prostate volume up to 75 cc (inclusive) documented by cross-sectional imaging (TRUS, MRI, etc.). Results from standard of care imaging may be accepted up to 6 months prior to Screening if the subject was not on 5-alpha reductase inhibitors (5ARIs) at that time
6. International Prostate Symptom Score (IPSS) ≥ 13
7. Maximum urinary flow rate (Qmax) of ≤ 15 mL/sec and ≥ 5 mL/sec (voided volume must be ≥ 125 mL)
8. Willing and able to complete all study visits including questionnaires at baseline and at follow-up visits

Exclusion Criteria:

1. History of prostate cancer or suspected, should be ruled out to the satisfaction of the PI by local standard of care methods within prior 6 months
2. Confirmed or suspected bladder cancer within the last 2 years
3. History of acute bacterial prostatitis within the last 2 years
4. Median lobe obstruction of the prostate as confirmed by cross-sectional imaging
5. PSA value > 10 ng/dl, ng/ml
6. Contraindicated for iTind or UroLift as determined by the PI
7. Neurogenic bladder and/or sphincter abnormalities due to Parkinson's disease, multiple sclerosis, cerebral vascular accident, diabetes or other neurological disorders that affect bladder function
8. Clinically significant bladder diverticulum
9. Diagnosed with urethral stricture, meatal stenosis, bladder neck contracture, rectal disease, artificial urinary sphincter, incompetent sphincter, urinary incontinence due to incompetent sphincter
10. Prior rectal surgery (other than hemorrhoidectomy) or history of rectal disease if the therapy may potentially cause injury to sites or previous rectal surgery (e.g., if a transrectal probe is used), pelvic radiotherapy or radical pelvic surgery, urinary diversion surgery, prostate surgery, balloon dilation, urethral stent implantation, laser prostatectomy, or any other invasive treatment to the prostate, or penile prosthesis that may prevent insertion of the iTind or UroLift device
11. An active urinary tract infection
12. Hematuria or cystolithiasis within the last 3 months
13. Prostate volume > 75 cc
14. Post-void residual volume (PVR) > 250 mL
15. Actively using catheterization or unable to void naturally
16. Unable to complete the required washout period for alpha blockers
17. Taking anti-platelet or anticoagulants (except low dose aspirin - 81 mg - 100 mg) within the last 7 days prior to randomization
18. Known or suspected allergy to nickel, titanium or polyester/polypropylene

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of all intraoperative and post-operative complications | 3 months
  Incidence of all intraoperative and post-operative complications (i.e., related to procedure and/or device) at 3 months

SECONDARY OUTCOMES:
Difference in change from baseline between iTind and UroLift groups in International Prostate Symptom Score (IPSS) | 1, 3, 6, 12, 24, 36, 48, and 60 months
  Difference in change of International Prostate Symptom Score (IPSS) from baseline between iTind and UroLift groups
Difference in change of QoL scores from baseline between iTind and UroLift | 1, 3, 6, 12, 24, 36, 48, and 60 months
  Difference in change of QoL scores from baseline between iTind and UroLift
Difference in rate of re-intervention | 1, 3, 6, 12, 18, 24, 36, 48, and 60 months
  Difference in rate of re-intervention between iTind and UroLift groups
Difference in reporting between iTind and UroLift groups | 1, 3, 6, 12, 18, 24, 36, 48, and 60 months
  Difference in reporting between iTind and UroLift groups in overall incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Chughtai, MD, Principal Investigator — Plainview Hospital; Neil Barber, MD, Principal Investigator — Frimley Park Hospital
Locations (18):
- United States (15):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Arizona Urology Specialists, Tucson, Arizona
  - Urology Associates of Central California, Fresno, California
  - Golden State Urology, Sacramento, California
  - NorthShore University Health System Research Institute, Evanston, Illinois
  - Southeast Louisiana Veterans Health Care System, New Orleans, Louisiana
  - Minnesota Urology, Woodbury, Minnesota
  - Adult & Pediatric Urology, Omaha, Nebraska
  - Pacific West Urology, Las Vegas, Nevada
  - Feinstein Institutes for Medical Research / Northwell Health, Syosset, New York
  - The Conrad Pearson Clinic, Germantown, Tennessee
  - Midtown Urology Associates, Austin, Texas
  - Houston Metro Urology, Houston, Texas
  - The Urology Place, San Antonio, Texas
  - Potomac Urology Center, Alexandria, Virginia
- United Kingdom (3):
  - Queen Margaret Hospital, Dunfermline
  - Frimley Park Hospital, London
  - Norfolk & Norwich University Hospital, Norwich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company website — https://www.itind.com/